CLINICAL TRIAL: NCT04424420
Title: Double Blinded Randomized Placebo Controlled Study on Mental Effects of Analgesic Drugs
Brief Title: Mental Effects of Analgesic Drugs: Paracetamol and Ibuprofen
Acronym: MEAD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Jürgen Brockmöller (Other)
Collaborators: University Hospital Ulm (Other)
Responsible Party: Sponsor-Investigator, Prof. Jürgen Brockmöller, Director, Institute of Clinical Pharmacology at Universitätsmedizin Göttingen, University of Göttingen
Organization: University of Göttingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018-004187-60
Record Dates: First submitted 2020-02-18; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Empathy
Keywords: Mental effects; Social Pain
MeSH Terms: interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective with placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracetamol (Experimental): Study phase 1 (single dosing): 1000 mg once. Study phase 2 (multiple dosing): 1000 mg twice daily for a minimum of 12 and a maximum of 14 days.
  Interventions: Drug: Paracetamol
- Ibuprofen (Active Comparator): Study phase 1 (single dosing): 800 mg once.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Study phase 1 (single dosing): Once. Study phase 2 (multiple dosing): Twice daily for a minimum of 12 and a maximum of 14 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Paracetamol — Paracetamol oral tablet
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Ibuprofen — Ibuprofen oral tablet
  Arms: Ibuprofen
Drug: Placebo oral tablet — Sugar pill manufactured to mimic the Paracetamol and Ibuprofen.
  Arms: Placebo

SUMMARY:
The objective of the present study is to study paracetamol effects on social pain and empathy under standardized international conditions (ICH-GCP) for planning, conduction and reporting of clinical pharmaceutical studies in humans. The study included MRI imaging of brain activity, analysis of genomic biomarkers potentially explaining interindividual variation. It is controversial whether the effects are of immediate nature or develop during a period of about 10 days. Therefore, the study is separated into two study phases. Single dosing (SD) is applied in study phase 1 and multiple-dosing (MD) in study phase 2. The study compares paracetamol with placebo and in the study phase 1 also with ibuprofen as analgetically active control.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to study.
2. Willingness to meet the study instructions and to co-operate with the study personal.
3. No clinically relevant pathological findings in any of the investigations at the screening visit; minor deviations of laboratory values from the normal range may be accepted if judged by the investigator to have no clinical relevance.
4. Body weight not less than 48 kg and body mass index (BMI) not less than 17 kg/m² and not greater than 32 kg/m².

Exclusion Criteria:

1. Pacemaker devices, implantable or external ones.
2. Involvement in the planning and conduct of the study (applies to staff directly employed at the study site / department).
3. Known pregnancy or lactation period.
4. History of alcohol and / or drug abuse and / or any abusive use of medicaments.
5. Any disease affecting liver or kidney or impairment of the liver or kidney-function.
6. History of severe hypersensitivity reactions, anaphylaxis, psychiatric or neurologic disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effect of paracetamol and ibuprofen on social pain and empathy | 8 hours
  Primary outcome is defined as the composite score of standardized emotional scenarios and the hurt feeling scale.
Effect of paracetamol on social pain and empathy | 14 days
  Primary outcome is defined as the composite score of standardized emotional scenarios and the hurt feeling scale.

SECONDARY OUTCOMES:
Psychological effects of paracetamol and ibuprofen | 8 hours
  Interindividual variation of analgesic effects measured using fMRI. MRI will be performed to reflect differences in brain activation by Psychometric test.
Pharmacokinetics effects of paracetamol and ibuprofen | 8 hours
  Blood samples for determination of study drug concentrations in plasma will be taken at different time-point. This will be used to calculate Maximum Plasma Concentration (Cmax).
Pharmacogenes roles in paracetamol and ibuprofen metabolism | 8 hours
  Genetic analysis of relevant genes responsible for paracetamol and ibuprofen Absorption, Distribution, Metabolism and Excretion (ADME).Healthy volunteers will provide a blood sample for molecular genetic analyses of the various candidate genes, e.g. drug transporters and metabolizing enzymes. This will shed light on the interindividual variation of analgesic effects.
Psychological effects of paracetamol | 14 days
  Interindividual variation of analgesic effects measured using fMRI. MRI will be performed to reflect differences in brain activation by Psychometric test.
Pharmacokinetics effects of paracetamol | 14 days
  Blood samples for determination of study drug concentrations in plasma will be taken at different time-point. This will be used to calculate Maximum Plasma Concentration (Cmax).
Pharmacogenes roles in paracetamol metabolism | 14 days
  Genetic analysis of relevant genes responsible for paracetamol Absorption, Distribution, Metabolism and Excretion (ADME). Healthy volunteers will provide a blood sample for molecular genetic analyses of the various candidate genes, e.g. drug transporters and metabolizing enzymes. This will shed light on the interindividual variation of analgesic effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Göttingen, Göttingen, Lower Saxony, Germany